CLINICAL TRIAL: NCT05411835
Title: Safety and Tolerability of Oral Ketones and Exercise Among Patients With Long-chain Fatty Acid Oxidation Disorders
Brief Title: Oral Ketones and Exercise Among Patients With Long-chain Fatty Acid Oxidation Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Melanie B Gillingham, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 23859
Record Dates: First submitted 2022-05-27; First posted 2022-06-09 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2022-10

CONDITIONS: Long-chain 3-hydroxyacyl-CoA Dehydrogenase Deficiency; Carnitine Palmitoyltransferase Deficiency 2; Very Long Chain Acyl Coa Dehydrogenase Deficiency; Trifunctional Protein Deficiency
MeSH Terms: conditions — Trifunctional Protein Deficiency With Myopathy And Neuropathy; Carnitine palmitoyl transferase 2 deficiency; VLCAD deficiency

STUDY DESIGN:
Intervention Model Description: Subjects with either CPT2, TFP, LCHAD or VLCAD deficiency will be randomized to receive a ketone beverage (see composition in Appendix A) or an isocaloric maltodextrin control beverage (see composition in Appendix A) before moderate intensity exercise. Twenty minutes after consuming the pre-exercise beverage, subjects will complete a moderate intensity treadmill exercise test for 45 minutes. After a washout period of 48 hours, subjects will repeat the exercise. During the 2nd exercise test subjects will crossover to the beverage not consumed during the 1st exercise study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sachets of the ketone or maltodextrin powder are coded and packaged identically. The bionutrition unit will prepare the beverage and maintain the randomization code and the code for the ketone and maltodextrin products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Ketogenic Supplement (Active Comparator): The Ketone pre-exercise beverage is a nutritional supplement. The supplement will be provided by Nestle as powered sachets to mix in water. It contains a mix of D-beta-hydroxybutyrate salts, flavors and stevia.
  Interventions: Dietary Supplement: Nutritional Ketone Supplement
- Isocaloric Placebo Supplement (Sham Comparator): The maltodextrin pre-exercise beverage is a nutritional supplement. The supplement will be provided by Nestle as powered sachets to mix in water. It contains an isocaloric amount of maltodextrin, flavors and stevia similar to the ketone beverage.
  Interventions: Dietary Supplement: Isocaloric Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Nutritional Ketone Supplement — Mix of sodium, calcium, and magnesium salts of D-beta-hydroxybutyrate with nicotinamide riboside chloride, flavors and stevia sweetener
  Other Names: NKS
  Arms: Nutrition Ketogenic Supplement
Dietary Supplement: Isocaloric Placebo Supplement — Maltodextrin with flavors and stevia sweetener
  Arms: Isocaloric Placebo Supplement

SUMMARY:
The purpose of the study is to determine if an oral ketone beverage is safe and well-tolerated during moderate intensity exercise in participants with long-chain fatty acid oxidation disorders and if it will raise blood ketones to levels similar to that reported among normal healthy subjects.

DETAILED DESCRIPTION:
Purpose: Subjects with long-chain fatty acid oxidation disorders (LC-FAOD) do not make ketones during fasting or with exercise. Ketones are an important alternative energy substrate during moderate exercise, sparing the oxidation of glucose and providing a source of ATP to the central nervous system and exercising muscle. Fatty acid oxidation in the liver is required to make ketones. Subjects with a LC-FAOD cannot generate ketones because of their block in fatty acid oxidation during exercise. Providing ketones in an oral ketone beverage may increase blood ketones with exercise to levels normally observed in humans.

Aim: To determine the safety and tolerability of an oral ketone beverage during moderate intensity exercise among subjects with a LC-FAOD compared to an isocaloric maltodextrin beverage, and to determine blood ketone concentrations.

Hypothesis: Oral consumption of a ketone beverage before moderate intensity exercise will be safe and well-tolerated, and will raise blood ketones among subjects with a LC-FAOD to concentrations similar to that reported in the literature among normal healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of VLCAD, LCHAD/TFP or CPT2 deficiency
* speak English
* willing to complete 2 moderate intensity exercise treadmills

Exclusion Criteria:

* subjects actively participating in another research study that prohibits their participation
* pregnant females
* subjects with diabetes or taking medications to treat diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Adverse Events- incidence | 2 hours after product intake
  Number of Adverse events
Adverse Events- type | 2 hours after product intake
  Description of Adverse events: categorical
Adverse Events- severity | 2 hours after product intake
  Severity of adverse event: grade 1-5
Adverse Events- causal relationship | 2 hours after product intake
  Yes/No related to product intake
Abdominal discomfort | 2 hours after product intake
  visual analogue scale (VAS) 0-10
Decreased appetite | 2 hours after product intake
  visual analogue scale (VAS) 0-10
Gastric reflux | 2 hours after product intake
  visual analogue scale (VAS) 0-10
Nausea | 2 hours after product intake
  visual analogue scale (VAS) 0-10
Diarrhea | 2 hours after product intake
  visual analogue scale (VAS) 0-10
Headache | 2 hours after product intake
  visual analogue scale (VAS) 0-10

SECONDARY OUTCOMES:
Blood Ketones | 20 minutes after moderate intensity exercise
  plasma beta-hydroxybutyrate concentration
Blood Creatine Kinase | 20 minutes after moderate intensity exercise
  plasma CK concentration
Blood Glucose | 20 minutes after moderate intensity exercise
  serum glucose
Blood Lactate | 20 minutes after moderate intensity exercise
  serum lactate concentration
Blood Pressure | peak 40 minute exercise
  diastolic BP
Blood Pressure | peak 40 minute exercise
  systolic BP
Perceived exertion | peak 40 minute exercise
  Borg scale 1-20
Respiratory Exchange Ratio | peak 40 minute exercise
  VCO2/VO2 0.7 - 1.0
Heart Rate | peak 40 minute exercise
  beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will be provided with creatine kinase lab test and body composition measurement. The results of their creatine kinase lab test will be placed in their medical record. Results of the study will be written in a published manuscript and summarized in a cover letter to be sent via mail or email to the participant after publication of the data.
Supporting Information: Study Protocol, ICF
Time Frame: The published manuscript will be available approximately 6-9 months after the conclusion of the study.
Access Criteria: not applicable. A reprint will be sent to participants.